CLINICAL TRIAL: NCT05719454
Title: Clinical Feasibility of a Novel Setup Algorithm for BackBeat Medical's Cardiac Neuromodulation Therapy (CNT) Pacing Signals
Brief Title: Novel Setup Algorithm for Cardiac Neuromodulation Therapy
Acronym: CS-10
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: BackBeat Medical Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CS-10 BBM NOV SA
Record Dates: First submitted 2023-01-09; First posted 2023-02-09 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Hypertension; Bradycardia
MeSH Terms: conditions — Hypertension; Bradycardia

STUDY DESIGN:
Intervention Model Description: All subjects will undergo in visits 4 and 5 two sessions to test two different setup CNT Algorithms. One version will favor atrial pacing. The order of the setup versions will alternate, whereby subjects will start with setup version 1 or setup version 2 Subjects will be sequentially assigned to Version 1 or 2 on alternating basis: first subject to Version 1, second to Version 2, third to Version 1, etc. hey will also undergo setup without the use of an algorithm, similar to the method used in the MODERATO II study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CNT Setup Algorithm Version 1 (Experimental): When performing the Setup Algorithm Version 1, each subject's blood pressure is measured with a standard cuff system while the BackBeat-CNT is activated, and system parameters are varied successively according to a specified sequence or based on the blood pressure measurements obtained during previous activations of BackBeat CNT, until the Setup Algorithm is complete. The parameter values as determined by the Setup Algorithm will constitute the programming of the Moderato IPG for the 24 hour activation following setup.
  Interventions: Device: CNT testing
- CNT Setup Algorithm Version 2 (Experimental): When performing the Setup Algorithm Version 1, each subject's blood pressure is measured with a standard cuff system while the BackBeat-CNT is activated, and system parameters are varied successively according to a specified sequence or based on the blood pressure measurements obtained during previous activations of BackBeat CNT, until the Setup Algorithm is complete. The parameter values as determined by the Setup Algorithm will constitute the programming of the Moderato IPG for the 24 hour activation following setup.
  Interventions: Device: CNT testing
- CNT therapy optimization without use of the Setup Algorithm (Other): For this optimization procedure, each subject's blood pressure is measured with a continuous blood pressure measurement system while the BackBeat-CNT is activated, and system parameters are varied according to a specified sequence until the desired blood pressure reduction is achieved. The parameter values that provide the desired blood pressure reduction will be recorded, for possible use by the investigator following trial completion
  Interventions: Device: CNT testing

INTERVENTIONS:
Device: CNT testing — The effect of CNT on blood pressure will be obtained throughout the year long follow up period.

SUMMARY:
After meeting all inclusion/exclusion criteria, subjects on standard pacing with the Moderato® Implantable Pulse Generator (IPG) will be subjected to two set-up sessions for the CNT algorithm: at week 4 and at week 6 post implant. At the end of these visits, subjects will undergo a 24 ambulatory blood pressure recording after which CNT will be automatically turned OFF and standard pacing will resume.

The ambulatory data will provide the basis for a lasting CNT programming by week 8. Follow up visits will be scheduled after 3, 6, and 12 months.

DETAILED DESCRIPTION:
This is a feasibility, pilot, interventional clinical study comparing the performance of CNT pacing signals delivered by Moderato® System using a new Setup Algorithm to the performance of the CNT pacing signals delivered by Moderato® System in a similar patient population in a previous multi-center, randomized, double blinded chronic trial (MODERATO II, described below).

Subjects meeting all eligibility criteria (detailed below) will receive a Moderato® IPG (Implantable Pulse Generator), either as a new implant or as a replacement to an existing pacemaker (visit 2). The subject will then be observed during the "Run-in Phase" for 30 days with the device programmed to deliver standard pacing therapy. During the "Run-In Phase", 3 weeks from implant (visit 3), the subjects will undergo a 24-hour Ambulatory Blood Pressure Measurement (ABPM). At the end of the "Run-in Phase" (4 weeks from implant at visit 4), eligibility for activation of CNT pacing signals will be re-established. Subjects eligibility will be determined following the result of the 24-hour ABPM conducted at week 3 from implant and office blood measurement at week 4 (inclusion criteria #5) and an assessment of change in ejection fraction from baseline using an echo measurement (exclusion criteria #5).

All subjects will undergo in visits 4 and 5 two sessions to test two different setup CNT Algorithms. One version will favor atrial pacing. The order of the setup versions will alternate, whereby subjects will start with setup version 1 or setup version 2 (see below). They will also undergo setup without the use of an algorithm, similar to the method used in the MODERATO II study.

After the "Run-In Phase", subjects meeting all eligibility criteria will undergo Setup Algorithm 1 (or 2). At the end of the visit, the Moderato® IPG will be programmed with the resulting CNT parameters to be delivered for 24 hours; after which the device will continue as a standard pacemaker with the pre-sets of the "Run-In Phase" period. Subjects will be fitted with 24 hour ABPM devices and sent home.

After two weeks (visit 5), subjects will return for the second setup visit. This time, subjects will undergo setup using the setup Algorithm version that was not used on them in the First Setup visit. They will also undergo setup without use of the algorithm, similar to the method used in the MODERATO II study. At the end of the second setup visit, the Moderato® IPG will be programmed using the resulting CNT parameters, to be delivered for 24 hours; after which the device will continue as a standard pacemaker with the pre-sets of the "Run-In Phase" period. Subjects will be fitted with 24 hour ABPM devices and sent home.

Subjects will return after two weeks for the trial CNT activation visit (visit 6). Based on the effect of the previous test CNT activations on blood pressure established by the two ABPM assessments, the investigator will decide whether to Continue CNT for the patient, with the parameters determined by the first or the second Setup Algorithm, or use the parameters established during setup without use of the algorithm.

Subjects will be further followed 3, 6 and 12 months post CNT activation (5, 8 and 14 months from implant) for changes in blood pressure and any adverse events (see study duration below).

At the end of the follow-up period, the treating physician will decide whether to leave CNT therapy on or off. Patient care will continue according to existing best practices.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years of age
* Subject requires implantation or replacement of a dual chamber pacemaker or requires an upgrade from a single chamber to a dual chamber pacemaker.
* Subject has stable (for prior 1 month) hypertension treatment with 1, 2 or 3 antihypertensive drugs, which is planned to be maintained without changes for a period of at least 2 months post implant.
* Subject has an office systolic blood pressure (oSBP) ≥140 and <180 mmHg
* At 4 weeks from device implant, subject has an average 24-Hour ambulatory systolic blood pressure (aSBP) ≥130 mmHg and <170 mmHg and an office blood pressure (oSBP) ≥140 and <180 mmHg.
* Subject is willing and able to comply with study visits and procedures
* Subject is willing to adhere to the prescribed baseline antihypertension medical regimen for the duration of the study.

Exclusion Criteria:

* 1. Subject has a known secondary cause of HTN (e.g. renal vascular disease, hyperthyroidism, hyperaldosterone and pheochromocytoma)
* Subject has permanent atrial fibrillation
* Subject has intermittent paroxysmal atrial fibrillation/flutter with significant burden (i.e., >10% atrial fibrillation/flutter beats if available.
* Subject has an ejection fraction <50%
* Subject has a drop of > 15% (absolute) in ejection fraction from baseline to week 4
* Subject has symptoms of heart failure, NYHA Class II or greater
* Subject has mitral regurgitation ≥2+, aortic stenosis with valve area <1.0 cm2 , or is expected to need a valve repair or replacement.
* Subject has a history of stroke or TIA within 12 months or any prior stroke with a residual neurological deficit (modified Rankin Score >2+)
* Subject experienced myocardial infarction (MI) within 3 months prior to enrolment
* Subject had a cardiovascular interventional procedure or cardiovascular surgery within 6 months prior to enrolment
* Subject has hypertrophic cardiomyopathy, restrictive cardiomyopathy or interventricular septal thickness ≥15 mm
* Subject is on dialysis
* Subject has estimated glomerular filtration rate (GFR) <30 ml/min/1.73m²
* Subject has significant (>50% occlusion of left or right carotid artery) carotid artery stenosis
* Subject has a history of clinically significant untreated ventricular tachyarrhythmia or has experienced sudden cardiac arrest
* Subject has an active device-based treatment for hypertension
* Subject has an existing active cardiac device or neurostimulator (e.g., ICD, spinal cord stimulator)
* Subject has Type I Diabetes
* Subject is a member of a vulnerable population (e.g., prisoners, pregnant or lactating women, mentally disabled)
* Subject has the possibility of becoming pregnant during the conduct of the study and is not willing to use a means of contraception during the study
* Subject cannot or is unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-21 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
CNT efficacy: Changes in average 24 hour systolic ambulatory blood pressure | up to 12 Month follow-up visit
  The change in the 24 hr blood pressure recording after each of the two set up sessions (week 4 and week 6) will be compared to the 24 hr ambulatory data of the control (week 3).
CNT safety: Incidence of device- and treatment-related adverse and serious adverse | up to 12 Month follow-up visit
  Incidence of device- and treatment-related adverse and serious adverse events during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Béla MERKELY, Prof. MD, Principal Investigator — Semmelweis University Heart and Vascular Center
Locations (7):
- Nemocnice Na Homolce (Na Homolce Hospital), Prague, Czechia
- Semmelweis University Heart and Vascular Center, Budapest, Hungary
- Poland (5):
  - Jagiellonian University Hospital, Krakow
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Poznan
  - Samodzielny Pub. Szpital Kliniczny nr 2 PUM, Szczecin
  - Publiczny Centralny Szpital, Warsaw
  - Silesian Center for Heart Diseases, Zabrze